CLINICAL TRIAL: NCT02230826
Title: Multicentric Observational PMCF Study to Evaluate Long-term Outcome, Performance and Safety of Implantable Devices in Hip Arthroplasty
Brief Title: Observational Study to Evaluate Long-Term Outcome in Hip Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: 1302-T-HIPLTO-RM
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Hip Replacement; Primary, Secondary or Post-traumatic Osteoarthrosis; Femur Head Necrosis; Congenital Dislocations; Primary and Revision Surgery
Keywords: Arthroplasty; Hip Replacement; Acetabular cup; Femoral stem
MeSH Terms: conditions — Neoplasm Metastasis; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Hip arthroplasty: Patients with Hip implants.

SUMMARY:
This long-term outcomes study is designed to collect safety and efficacy data on designated, commercially available, hip arthroplasty products.

DETAILED DESCRIPTION:
Outcome data collected from this study will be used for Post Market Surveillance (PMS) and Clinical Evaluations on Corin hip devices and will support peer-reviewed publications on products performance and safety at long term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman >18 years
* Subjects with indication of arthroplasty surgery with Corin hip devices which are under assessment as part of this PMCF study
* Subjects who agreed for study participation.

Exclusion Criteria:

* Subjects with existing tumour and/or particularly high surgical risk-
* Subjects with anaesthetic risk class IV or higher
* Subjects under guardianship and/or unable to follow procedures or matters related to the study (examples: Illiterate, recent psychotic or mania disorders and / or inability to comply with usual follow-up visits.)
* Contraindications for arthroplasty with a Corin hip devices as per product IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients with a partial or total hip replacement (Corin implants)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-05; Primary Completion 2034-12 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of long-term outcome after hip arthroplasty with Corin implants. | At 10 years
  Implants revision rate at 10-year FU hip arthroplasty

SECONDARY OUTCOMES:
Evaluation of long-term outcome after hip arthroplasty with Corin implants at 15 and 20-year FU. | at 15- and 20-year
  Implants revision rate at 15- and 20-year FU.
Evaluation of clinical performance of Corin hip implants | starting intraoperatively up to 20-year FU
  Change of Patient Reported Outcome Measures (PROMs)
Evaluation of Safety of Corin hip implants | starting intraoperatively up to 20-year FU
  Number, severity and causal relationship of procedure or implant-related Adverse Events
Radiological evaluation of positioning and osteointegration of Corin hip implants. | starting intraoperatively up to 20-year FU
  Number, thickness and location of radiolucent lines, osteolysis and heterotopic ossifications reported via radiological evaluation
Evaluation of patient quality of life | starting intraoperatively up to 20-year FU
  Improvement of quality of life via EQ-5D-5L scores.
Evaluation of patient satisfaction following surgery | 3 months ; 2.5-year; 6, 11, 15, 20-year visits
  Improvement of patient's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Goulven Rochcongar, MD, Study Chair — University Hospital, Caen
Locations (13):
- France (13):
  - CHU de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - clinique Oxford Cannes, Cannes
  - CH Dunkerque, Dunkirk
  - Polyclinique Henin Beaumont, Hénin-Beaumont
  - CHU de Nice, Nice
  - Centre Hospitalier Régionnal d'Orléans - Site La Source, Orléans
  - Clinique Arago, Paris
  - Hôpital de la Croix Saint-Simon, Paris
  - Hopital privé Saint-Martin, Pessac
  - Hôpital Provo, Roubaix
  - Polyclinique St Georges de Didonne, Saint-Georges-de-Didonne
  - Médipôle Garonne, Toulouse
  - Hôpital Jean Bernard, Valenciennes